CLINICAL TRIAL: NCT01469377
Title: A Double-Blind, Placebo-Controlled Study of Cariprazine (RGH-188) as Adjunctive Therapy in Major Depressive Disorder
Brief Title: Safety and Efficacy of Cariprazine as an Adjunctive to Antidepressant Therapy in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGH-MD-75
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo orally once a day for 8 weeks. Each participant continued to take the same dose of antidepressant therapy (bupropion, citalopram, desvenlafaxine, duloxetine, escitalopram, fluoxetine, sertraline, venlafaxine, or vilazodone) the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Placebo
- Cariprazine 1-2 mg (Experimental): Participants received cariprazine orally once a day for 8 weeks. Participants received cariprazine 0.5 mg on Days 1 and 2 and 1.0 mg on Days 3-7. At the investigator's discretion dose levels could be increased during Week 2. Dose levels allowed during Week 2 were 1.0 or 1.5 mg. A second dose increase was allowed starting at Week 3. Dose levels allowed during Week 3 and the remainder of the treatment period were 1.0, 1.5, or 2.0 mg. Each participant continued to take the same dose of antidepressant therapy (bupropion, citalopram, desvenlafaxine, duloxetine, escitalopram, fluoxetine, sertraline, venlafaxine, or vilazodone) the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Cariprazine
- Cariprazine 2-4.5 mg (Experimental): Participants received cariprazine orally once a day for 8 weeks. Participants received cariprazine 0.5 mg on Days 1 and 2, 1.0 mg on Day 3, 1.5 mg on Day 4, and 2.0 mg on Days 5-7. At the investigator's discretion dose levels could be increased during Week 2. Dose levels allowed during Week 2 were 2.0 or 3.0 mg. A second dose increase was allowed starting at Week 3. Dose levels allowed during Week 3 and the remainder of the treatment period were 2.0, 3.0, or 4.5 mg. Each participant continued to take the same dose of antidepressant therapy (bupropion, citalopram, desvenlafaxine, duloxetine, escitalopram, fluoxetine, sertraline, venlafaxine, or vilazodone) the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Placebo — Placebo was supplied in capsules
  Arms: Placebo
Drug: Cariprazine — Cariprazine was supplied in capsules.
  Arms: Cariprazine 1-2 mg; Cariprazine 2-4.5 mg

SUMMARY:
An outpatient study to evaluate the safety and efficacy of cariprazine as adjunct to antidepressant therapy (ADT) in participants with major depressive disorder (MDD) who have an inadequate response to ADT alone. This clinical study compared cariprazine + ADT with placebo + ADT in outpatients with a diagnosis of MDD and an inadequate response to ADT. The study consisted of approximately 2 weeks of screening and washout followed by 8 weeks of double-blind treatment followed by a 1 week safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 to 65 years of age, inclusive.
* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for moderate to severe major depressive disorder (MDD).
* Current major depressive episode of at least 8 weeks and not exceeding 24 months in duration.
* Ongoing inadequate response to protocol allowed antidepressant therapy (ADT).

Exclusion Criteria:

* Principal DSM-IV-TR-based diagnosis of an axis I disorder, other than MDD,
* Women who are pregnant, or planning to become pregnant or breastfeed during the study or not practicing reliable contraception that will continue through out the study.
* History of meeting DSM-IV-TR criteria for:

  1. Depressive episode with psychotic or catatonic features.
  2. Manic, hypomanic or mixed episode, including bipolar disorder and substance induced manic, hypomanic or mixed episode.
  3. Schizophrenia, schizoaffective, or other psychotic disorder.
  4. Obsessive-compulsive disorder.
  5. Bulimia or anorexia nervosa.
  6. Dementia, amnesic, or other cognitive disorder.
  7. Mental retardation.
* Participants considered a suicide risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2011-12-15 (Actual); Primary Completion 2013-12-12 (Actual); Study Completion 2013-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, MD, Study Director — Allergan
Locations (72):
- United States (39):
  - Forest Investigative Site 077, Garden Grove, California
  - Forest Investigative Site 019, National City, California
  - Forest Investigative Site 039, Oceanside, California
  - Forest Investigative Site 015, Orange, California
  - Forest Investigative Site 050, Orange, California
  - Forest Investigative Site 008, Redlands, California
  - Forest Investigative Site 066, Sherman Oaks, California
  - Forest Investigative Site 063, Gainesville, Florida
  - Forest Investigative Site 029, Jacksonville, Florida
  - Forest Investigative Site 012, Kissimmee, Florida
  - Forest Investigative Site 023, Miami, Florida
  - Forest Investigative Site 026, Orlando, Florida
  - Forest Investigative Site 062, Atlanta, Georgia
  - Forest Investigative Site 065, Smyrna, Georgia
  - Forest Investigative Site 074, Prairie Village, Kansas
  - Forest Investigative Site 040, Flowood, Mississippi
  - Forest Investigative Site 068, Creve Coeur, Missouri
  - Forest Investigative Site 061, Cherry Hill, New Jersey
  - Forest Investigative Site 038, Marlton, New Jersey
  - Forest Investigative Site 030, Albuquerque, New Mexico
  - Forest Investigative Site 076, Brooklyn, New York
  - Forest Investigative Site 037, Mount Kisco, New York
  - Forest Investigative Site 067, New York, New York
  - Forest Investigative Site 049, New York, New York
  - Forest Investigative Site 047, Canton, Ohio
  - Forest Investigative Site 021, Dayton, Ohio
  - Forest Investigative Site 022, Portland, Oregon
  - Forest Investigative Site 027, Salem, Oregon
  - Forest Investigative Site 069, Bridgeville, Pennsylvania
  - Forest Investigative Site 025, Philadelphia, Pennsylvania
  - Forest Investigative Site 031, Reading, Pennsylvania
  - Forest Investigative Site 048, Memphis, Tennessee
  - Forest Investigative Site 024, Austin, Texas
  - Forest Investigative Site 020, Dallas, Texas
  - Forest Investigative Site 070, Houston, Texas
  - Forest Investigative Site 080, San Antonio, Texas
  - Forest Investigative Site 028, Salt Lake City, Utah
  - Forest Investigative Site 032, Bellevue, Washington
  - Forest Investigative Site 034, Kirkland, Washington
- Estonia (8):
  - Forest Investigative Site 203, Tallinn
  - Forest Investigative Site 201, Tallinn
  - Forest Investigative Site 206, Tallinn
  - Forest Investigative Site 205, Tallinn
  - Forest Investigative Site 204, Tartu
  - Forest Investigative Site 208, Tartu
  - Forest Investigative Site 207, Tartu
  - Forest Investigative Site 202, Võru
- Finland (7):
  - Forest Investigative Site 301, Helsinki
  - Forest Investigative Site 302, Helsinki
  - Forest Investigative Site 304, Helsinki
  - Forest Investigative Site 303, Helsinki
  - Forest Investigative Site 305, Kuopio
  - Forest Investigative Site 308, Oulu
  - Forest Investigative Site 307, Pori
- Slovakia (7):
  - Forest Investigative Site 602, Banská Štiavnica
  - Forest Investigative Site 603, Bardejov
  - Forest Investigative Site 604, Bratislava
  - Forest Investigative Site 606, Bratislava
  - Forest Investigative Site 601, Michalovce
  - Forest Investigative Site 605, Rimavská Sobota
  - Forest Investigative Site 607, Rimavská Sobota
- Sweden (3):
  - Forest Investigative Site 803, Lund
  - Forest Investigative Site 802, Malmo
  - Forest Investigative Site 801, Stockholm
- Ukraine (8):
  - Forest Investigative Site 705, Stepanivka, Kherson Oblast
  - Forest Investigative Site 703, Kharkiv
  - Forest Investigative Site 704, Kharkiv
  - Forest Investigative Site 702, Kyiv
  - Forest Investigative Site 701, Kyiv
  - Forest Investigative Site 710, Luhansk
  - Forest Investigative Site 709, Odesa
  - Forest Investigative Site 706, Vinnytsia

REFERENCES:
- [Derived] Durgam S, Earley W, Guo H, Li D, Nemeth G, Laszlovszky I, Fava M, Montgomery SA. Efficacy and safety of adjunctive cariprazine in inadequate responders to antidepressants: a randomized, double-blind, placebo-controlled study in adult patients with major depressive disorder. J Clin Psychiatry. 2016 Mar;77(3):371-8. doi: 10.4088/JCP.15m10070. PMID 27046309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Cariprazine 1-2 mg | Cariprazine 2-4.5 mg
Started | 269 | 274 | 276
Completed | 234 | 226 | 210
Not Completed | 35 | 48 | 66
Not completed — Protocol Deviation | 7 | 10 | 10
Not completed — Lost to Follow-up | 3 | 2 | 5
Not completed — Withdrawal of Consent | 12 | 14 | 15
Not completed — Adverse Event | 8 | 18 | 36
Not completed — Insufficient Therapeutic Response | 3 | 4 | 0
Not completed — Other Miscellaneous Reasons | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all subjects in the Randomized Population who received at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine 1-2 mg | Cariprazine 2-4.5 mg | Total
Number analyzed (Participants) | 266 | 273 | 273 | 812
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.6) | 45.5 (11.9) | 45.1 (11.4) | 45.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 187 | 201 | 578
  Male | 76 | 86 | 72 | 234
Race/Ethnicity, Customized [Number; unit: participants]
  White | 230 | 234 | 242 | 706
  All other races | 36 | 39 | 31 | 106
  Black or African American | 32 | 31 | 24 | 87
  Asian | 1 | 4 | 4 | 9
  American Indian or Alaska Native | 2 | 1 | 1 | 4
  Other | 1 | 3 | 2 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14 | 17 | 22 | 53
  Not Hispanic or Latino | 252 | 256 | 251 | 759
Weight [Mean (Standard Deviation); unit: kg] | 81.53 (16.19) | 79.69 (16.31) | 82.17 (17.37) | 81.13 (16.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.93 (5.09) | 28.21 (5.51) | 29.05 (5.59) | 28.73 (5.41)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 94.32 (13.44) | 93.36 (14.20) | 94.91 (14.66) | 94.20 (14.12)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Week 8
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Time Frame: Baseline to Week 8
Population: Intent-to-treat population consisted of all patients in the Safety Population who had at least 1 post-baseline assessment of the MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Cariprazine 1-2 mg | Cariprazine 2-4.5 mg
Number analyzed (Participants) | 264 | 273 | 271
Units on a scale | -12.5 (0.5) | -13.4 (0.5) | -14.6 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1-2 mg; Test type: Superiority; p = 0.2404, Mixed-effect model for repeated measures — p-values were from an mixed-effects model for repeated measures with treatment group, pooled study center, visit, and treatment-group-by-visit interaction as fixed effects and the baseline value and baseline value-by-visit interaction as covariates; p-values were adjusted for multiple comparisons using the matched parallel gate-keeping procedure; Least squares mean difference = -0.9, 95% CI 2-sided [-2.4 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 2-4.5 mg; Test type: Superiority; p = 0.0114, Mixed-effect model for repeated measures — [p-value comment as in outcome 1, analysis 1]; p-values were adjusted for multiple comparisons using the matched parallel gate-keeping procedure; Least squares mean difference = -2.2, 95% CI 2-sided [-3.7 to -0.6]

2. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The SDS measures an individual's perception of the extent to which his or her emotional symptoms are disrupting his or her functioning in 3 domains, work/school, social life/leisure activities, and family life/home responsibilities. The participant is asked to rate the degree to which their functioning is impaired on an 11-point scale, ranging from 0 (not at all) to 10 (extremely). Scores of 0 to 3 indicate mild functional impairment, 4 to 6 indicate moderate functional impairment, and 7 to 9 indicate marked functional impairment. The scores for the 3 domains are summed into a total score that ranges from 0 (unimpaired) to 30 (highly impaired). A higher score indicates greater impairment. A negative change score indicates improvement.
Time Frame: Baseline to Week 8
Population: Intent-to-treat population consisted of all patients in the Safety Population who had at least 1 post-baseline assessment of the MADRS total score. Only participants with scores for all 3 domains were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Cariprazine 1-2 mg | Cariprazine 2-4.5 mg
Number analyzed (Participants) | 264 | 273 | 271
Units on a scale | -6.6 (0.5) | -7.7 (0.5) | -8.0 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1-2 mg; Test type: Superiority; p = 0.2404, Mixed-effect model for repeated measures — [p-value comment as in outcome 1, analysis 1]; p-values were adjusted for multiple comparisons using the matched parallel gate-keeping procedure; Least squares mean difference = -1.1, 95% CI 2-sided [-2.5 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 2-4.5 mg; Test type: Superiority; p = 0.1140, Mixed-effect model for repeated measures — [p-value comment as in outcome 1, analysis 1]; p-values were adjusted for multiple comparisons using the matched parallel gate-keeping procedure; Least squares mean difference = -1.4, 95% CI 2-sided [-2.8 to 0.0]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected and recorded from the time the participant signs the informed consent form until 30 days after the last dose of treatment.
Description: Safety population: All randomized participants who received at least 1 dose of treatment.
Arm/Group | Placebo | Cariprazine 1-2 mg | Cariprazine 2-4.5 mg
All-Cause Mortality (participants affected / at risk) | 0/266 | 0/273 | 0/273
Serious Adverse Events (participants affected / at risk) | 1/266 | 0/273 | 3/273
Other Adverse Events (participants affected / at risk) | 102/266 | 121/273 | 179/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=266) | Cariprazine 1-2 mg (N=273) | Cariprazine 2-4.5 mg (N=273)
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Myocardial ischemia (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=266) | Cariprazine 1-2 mg (N=273) | Cariprazine 2-4.5 mg (N=273)
Constipation (Gastrointestinal disorders) | 5 | 6 | 14
Diarrhoea (Gastrointestinal disorders) | 14 | 8 | 8
Dry mouth (Gastrointestinal disorders) | 7 | 14 | 10
Nausea (Gastrointestinal disorders) | 13 | 19 | 35
Fatigue (General disorders) | 11 | 18 | 27
Increased appetite (Metabolism and nutrition disorders) | 4 | 5 | 14
Akathisia (Nervous system disorders) | 6 | 18 | 61
Dizziness (Nervous system disorders) | 7 | 10 | 14
Headache (Nervous system disorders) | 36 | 24 | 24
Somnolence (Nervous system disorders) | 14 | 24 | 27
Tremor (Nervous system disorders) | 4 | 13 | 21
Insomnia (Psychiatric disorders) | 17 | 27 | 38
Restlessness (Psychiatric disorders) | 7 | 22 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.